CLINICAL TRIAL: NCT05412238
Title: Formulation and Production of Macro- and Micronutrient Sachets for Home Fortification and Evaluation of Their Efficacy on Pregnant Mothers and Children Aged 6-60 Months in Sistan Baloochestan
Brief Title: Formulation and Evaluation of the Efficacy of Macro- and Micronutrient Sachets on Pregnant Mothers and Children Aged 6-60 Months
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Tirang R. Neyestani, Ph.D., Prof., National Nutrition and Food Technology Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 27
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Pregnancy; Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pregnant women receiving fortification sachets (Experimental): pregnant women receive daily fortified sachets containing micro-and macronutrients for 6-9 months
  Interventions: Dietary Supplement: micro-and macro-nutrients fortified sachets
- 6-24 months old children receiving fortification sachets (Experimental): 6-24 months old children receiv daily fortified sachets containing micro-and macronutrients for 6-9 months
  Interventions: Dietary Supplement: micro-and macro-nutrients fortified sachets
- 2-5 years old children receiving fortification sachets (Experimental): 2-5 years old children receive daily fortified sachets containing micro-and macronutrients for 6-9 months
  Interventions: Dietary Supplement: micro-and macro-nutrients fortified sachets

INTERVENTIONS:
Dietary Supplement: micro-and macro-nutrients fortified sachets — Every subject receives daily fortified sachets containing micro-and macronutrients for 6-9 months

SUMMARY:
The aim of the present study is formulation and production of sachets containing macronutrients and micronutrients to enrich food at home and evaluate its effectiveness on pregnant mothers and children aged 6 to 60 months living in Sistan and Baluchestan province

DETAILED DESCRIPTION:
This study is conducted in three steps. At first, fortification sachets are formulated and produced in accordance with international recommendations for micronutrients (vitamins A, D, zinc, and iron) and macronutrients for use in normal home conditions. In the second step, efficacy of fortified sachets are evaluate in three subgroups including pregnant mothers, 6-24 months and 2-5 years old children. Nutritional, anthropometrical and biochemical indices are evaluated at the beginning and after 6-9 months intervention. At the third step, costs and cost-effectiveness of the intervention in each of the studied groups in comparison with the usual program for that age group in the health care system of the country is determined.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women

   * being in the first trimester of pregnancy
   * free of chronic diseases before pregnancy
   * no intention to change residence until delivery
2. Children 6 to 23 months

   * age 6 to 7 months
   * no intention to change residence or migrate in the next 12 months
   * free of acute or chronic illness
3. Children 2 to 5 years (60-24 months)

   * age 24 to 48 months
   * no intention to change residence or migrate in the next 6-12 months
   * free of acute or chronic diseases

Exclusion Criteria:

1. Pregnant women

   * premature termination of pregnancy
   * change of residence before delivery
2. Children 6 to 23 months

   -change of residence before delivery
3. Children 2 to 5 years (60-24 months) -change of residence before delivery

Ages: 6 Months to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Weight gain during pregnancy | 6-9 months
  Weight difference at the beginning and end of pregnancy
Birth weight | 6-9 months
  Measured weight (kg) at the first day of life
Weight for age | 6-9 months
  Measured weight (kg) in a specific age (year)
Weight for height | 6-9 months
  The ratio of weight (kg) to height(m)

SECONDARY OUTCOMES:
25-hydroxyvitamin D (nmol/L) | 6-9 months
  Fasting serum 25-hydroxyvitamin D level
Hemoglobin (g/dL) | 6-9 months
  Blood hemoglobin level
Serum ferritin (ng/mL) | 6-9 months
  Fasting serum ferritin level
Serum zinc (microg/dL) | 6-9 month
  Fasting serum zinc level
Serum retinol (micromol/L) | 6-9 months
  Fasting serum retinol level
Serum folate (ng/mL) | 6-9 months
  Fasting serum folate level
Serum B12 (pg/mL) | 6-9 months
  Fasting serum B12 level
Apgar score | 6-9 months
  The Apgar score is a quick evaluation of one minute and five minutes after birth which tests the birthing process and readiness of newborn to meet the world without additional medical assistance

CONTACTS AND LOCATIONS:
Overall Officials: Tirang R. Neyestani, PhD, Study Chair — NationalNFTI, SBMU, Tehran, Iran
Locations (1):
- Laboratory of Nutrition Research, National Nutrition and Food Technology Research Institute (NNFTRI) and Faculty of Nutrition Science and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran, Iran, Tehran, Iran